CLINICAL TRIAL: NCT00447200
Title: Study of the Natural Variation in Strokevolume, and Investigation in the Number of Cycles Necessary to Find a 10% Strokevolume Variation Using Esophageal Doppler
Brief Title: Study of the Natural Variation in Strokevolume
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: Validation of cycles
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Last update posted 2007-10-15 (Estimated); Status verified 2007-10

CONDITIONS: Stroke Volume Variation
Keywords: Stroke volume; SV variation; Esophagus Doppler; Goal Directed Therapy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Esophagus Doppler monitoring
Procedure: Fluid optimization

SUMMARY:
We would like to investigate the natural variation in the strokevolume of the heart. At the same time we would like to find out the minimal number of heart cycles necessary to discover a 10% increase in strokevolume, after a fluid bolus of 200ml Voluven, when using Esophageal Doppler.

DETAILED DESCRIPTION:
We would like to investigate the natural variation in the strokevolume(SV) of the heart. At the same time we would like to find out the minimal number of heart cycles necessary to discover a 10% increase in SV, after a fluid bolus of 200ml Voluven, when using Esophageal Doppler.

Also we will compare the variation in SV both before and after the patients have been fluid optimized, using an algorithm of 10% increase in SV in order to receive another fluid bolus. The equipment used, will be the CardioQ from Deltex medical.

ELIGIBILITY:
Inclusion Criteria:

* Planned abdominal surgery

Exclusion Criteria:

* Oesophageal pathology,
* Age >90 yr or <18 yr,
* Alcohol abuse,
* Aneurism in thoracic aorta

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-03; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Strokevolume variation before fluid optimization
Strokevolume variation after fluid optimization
Number of cycles needed in order to detect a 10% strokevolume increase after fluid bolus of 200ml Voluven.

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Jorgensen, M.S, Principal Investigator — Dept of anesthesia 2041, ABD centre, Rigshospitalet, Blegdamsvej
Locations (1):
- Rigshospitalet, Copenhagen, Region Sjælland, Denmark